CLINICAL TRIAL: NCT03743168
Title: The Acute Effects of Intermittent Versus Continuous Bilateral Ankle Plantar Flexors Static Stretching on Postural Sway and Plantar Pressures During Standing
Brief Title: Static Stretching on Postural Sway and Plantar Pressures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Static-Stretching
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Muscle Stretching Exercise; Postural Balance; Stabilometry; Platform

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent stretching protocol (Experimental): Intermittent stretching protocol including five sets at 1 minute and 15 second rest.
  Interventions: Other: Intermittent stretching protocol
- Continuous stretch (Experimental): 2 minutes continuous stretch
  Interventions: Other: Continuous stretch

INTERVENTIONS:
Other: Intermittent stretching protocol — Intermittent stretching protocol of five sets of 1 minute and15 second rest
  Arms: Intermittent stretching protocol
Other: Continuous stretch — 2 minutes continuous stretch
  Arms: Continuous stretch

SUMMARY:
Risk for falls has been associated with falls efficacy and postural balance. The objective was to compare the effects on the footprint and the stabilometry of the continuous stretch and the intermittent. Subjects were randomly assigned to an intermittent stretching protocol group or continuous stretch group both of them loading passive plantar flexor stretching. Static footprint and stabilometry were measured before and after both protocols.

ELIGIBILITY:
Inclusion Criteria:

* Non-trained individuals
* Healthy subjects

Exclusion Criteria:

* Previous surgery on the lower extremities
* Injuries
* Musculoskeletal conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Foot plantar pressure | Change from foot plantar pressure at 2 minutes
  Maximum foot plantar pressure measured as K Pa

CONTACTS AND LOCATIONS:
Locations (1):
- Ricardo Becerro de Bengoa Vallejo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Jimenez EM, Losa-Iglesias ME, Gonzalez-Martin S, Lopez-Lopez D, Roca-Dols A, Rodriguez-Sanz D, Becerro-de-Bengoa-Vallejo R, Calvo-Lobo C. A 120-second stretch improves postural control and plantar pressure: quasi-experimental study. Sao Paulo Med J. 2022 May-Jun;140(3):341-348. doi: 10.1590/1516-3180.2021.0255.23072021. PMID 35508003